CLINICAL TRIAL: NCT04447495
Title: Self-sampling for the Study of COVID-19
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Juan C. Felix, MD, Professor, Medical College of Wisconsin
Other Study IDs: 20-001
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — A dry swab will be collected from two of the three iAMP® self-sample sites - mid-turbinate and anterior nares.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SARS-CoV-2 positive: We will enroll patients within a larger clinical validation study of the iAMP® test against the gold standard (the CDC-recommended test) until we have prospectively collected a total of 100 positive cases.
  Interventions: Diagnostic Test: iAMP test
- Controls: Current SARS-CoV-2 positivity in the region is approximately 20%, therefore, approximately 400 negative control samples will be needed.
  Interventions: Diagnostic Test: iAMP test

INTERVENTIONS:
Diagnostic Test: iAMP test — The low-cost Atila BioSystems iAMP® COVID-19 Detection kit consists of a reaction buffer mix, primer mix, three sample buffer components, a positive and negative control, nasopharyngeal swabs, and sample collection vials. Each kit is suitable for 100 tests.

SUMMARY:
This study will evaluate the feasibility of self-sampling with the iAMP® COVID-19 Detection Kit (Atila BioSystems, Mountain View, CA), a new, low-cost SARS-CoV-2 test that does not require RNA extraction. The investigators will compare the sensitivity and specificity of the iAMP® assay on self-sampled mid-turbinate, anterior nares, and saliva swabs against the gold standard, a nucleic acid amplification testing assay on a clinician-collected nasopharyngeal swab.

DETAILED DESCRIPTION:
3.1.1 Study population: The investigators will enroll patients within a larger clinical validation study of the iAMP® test against the gold standard (the CDC-recommended test) until we have prospectively collected a total of 100 positive cases. Current positivity in the region is approximately 20%, therefore, approximately 500 samples will be needed. Inclusion criteria are as follows: Patients older than 18 presenting for COVID-19 testing, able to tolerate nasopharyngeal swabs, and able to follow instructions for self-collection. Exclusion criteria are as follows: unable or unwilling to provide informed consent and/or reliable contact information.

3.1.2 Clinical visit: Symptomatic patients will be approached by a study provider wearing PPE. The study will be explained and if the patient agrees, they will be consented. Patients will be allowed to consent for just the two nasopharyngeal swabs or for all five swabs. After consent, each patient will undergo testing with simultaneous placement of two nasopharyngeal swabs by a clinician for the large-scale clinical validation. One will be stored dry in a tube and one will be placed in viral collection medium. Patients who consent to the self-sampling study will be taken to a private area for collection of three different samples. After receiving written instructions and watching a short instructional video, the mid-turbinate sample will be collected by the patient under the supervision of a clinician. The clinician will then leave and the patient will self-collect samples from the anterior nares and saliva. All samples will be stored dry. When the patient returns the samples to the research coordinator, they will be asked about any side effects or adverse events from the mid-turbinate sample.

3.1.3 Laboratory testing: A dry swab will be collected from two of the three iAMP® self-sample sites - mid-turbinate and anterior nares - and placed into a vial with the proprietary buffer (hereafter referred to as Sample Buffer A). For saliva, a sterile collection cup will be used for the sample collection, and Sample Buffer A will be added directly to the sterile collection cup. Each of the three samples with the added Sample Buffer A will incubate at room temperature for 15 minutes. A proprietary multiplex mixture (master mix) will be prepared in a test tube and 10 microliters of the sample from the vial (mid turbinate and nares) or cup (saliva) will be added to the test tube. The test tube will then be placed into the RT-PCR machine and run to completion of the assay. The assay will be resulted as either positive, negative or invalid (test to be repeated) and the result compared to the anonymized result of the nasopharyngeal test run with the CDC recommended NAAT assay.

Instructions for subjects on how to correctly collect the swabs from each site. [Cotton swabs should be flocked and tapered].

Mid-turbinate:

* Wash and dry hands thoroughly
* Take a sterile cotton swab and hold it by the stem in your dominant hand
* Open the empty iAMP collection vial and hold it in the other hand
* Tilt your head back so chin is roughly parallel to ground (~70º)
* Insert the cotton swab to the mark on the stem (one inch, or ~2 cm) and rotate the cotton swab completely (360º) 3 times.
* Remove the swab and without touching the cotton tip, repeat the process on the other side with the same cotton swab
* Remove the swab from the nose, do not touch the cotton tip, and place the swab, cotton tip first, into the vial
* Break off the upper stem of the cotton swab
* Replace the cap onto the vial, closing it securely
* Give the closed vial to the research personnel

Anterior nares:

* Wash and dry hands thoroughly
* Take a sterile cotton swab and hold it by the stem in your dominant hand
* Open the empty iAMP® collection vial and hold it in the other hand
* Insert the cotton swab into one nostril just until the cotton tip is no longer visible (~0.5 inches, or 1 cm)
* Rotate it inside the nose completely (360º) 3 times and leave it in place for 10-15 seconds
* Remove the swab and without touching the cotton tip, repeat the process in the other nostril, again inserting the cotton swab only until the cotton tip is no longer visible, rotating it 3 times and leaving it in place for 10-15 seconds
* Remove the swab, do not touch the cotton tip, and place the swab, cotton tip first, into the vial
* Break off the upper stem of the cotton swab
* Replace the cap onto the vial, closing it securely
* Give the closed vial to the research personnel

Saliva:

* Do not eat, drink, smoke or chew gum within 30 minutes of the collection
* Take a sterile urine cup and spit repeatedly into it until there is 2-3 milliliters of liquid (excluding bubbles). See image below for example of amount of saliva needed
* Keep inside of cup sterile by NOT placing anything (fingers, objects, etc) into the cup
* Once adequate amount of saliva collected, place the cap onto the top of the cup and close it securely
* Give closed cup to research personnel

3.1.4 Statistical justification Assuming 20% of specimens tested with the NAAT assay will be COVID-19 positive, a study of 500 consecutive specimens will yield 100 COVID-19 cases detected by the NAAT assay. This study will be able to estimate the 95% confidence interval (CI) for sensitivity and specificity indicated in the table below for true sensitivity and specificity ranging from 50% to 95%. The precision improves the farther the sensitivity and specificity differ from 50%.

Table 1: 95% confidence intervals for detecting sensitivity and specificity True Sensitivity Sensitivity 95% CI True Specificity Specificity 95% CI 50% 39.8% - 60.2% 50% 45.0% - 55.0% 70% 60.0% - 78.8% 70% 65.2% - 74.5% 90% 82.4% - 95.1% 90% 86.6% - 92.8% 95% 88.7% - 98.4% 95% 92.3% - 96.9%

3.1.5 Risks/Safety The only risk of this study is the additional exposure of the laboratory personnel performing the assay. All laboratorians involved are trained in handling infectious agents such as COVID-19. All standard precautions will be used for the handling of the specimens including aliquoting samples in a Biosafety hood and the use of Personal Protective Equipment. Patient confidentiality will be assured by the anonymizing of patient samples as previously approved by the MCW IRB.

3.1.6 Analysis. Sensitivity and specificity will be estimated for each iAMP® test as well as corresponding 95% exact confidence intervals using the NAAT assay as the reference standard.

3.1.7 Potential Clinical Limitations

1. Alternative anatomic sites will have lower sensitivity than nasopharyngeal swabs. It is possible that the self-collected swabs will have significantly lower sensitivity than nasopharyngeal swabs. This is unlikely to be the case because viral load with this novel virus is very high
2. Subjects may refuse to have multiple swabs taken. Patients may refuse to give 5 samples. Since the self-collected sites are unlikely to cause discomfort we expect that most participants will agree to study participation. Even if many patients do not agree to participate there are 700 patients per day presenting with symptoms which a large pool of potential participants which will make it feasible to reach our goal. The investigators may need to continue enrollment until there are 100 self-collected COVID-19 + subjects if some subjects refuse additional tests.

3.2 Specific Aim 2. Evaluate the incidence of adverse events in a self-collected mid-turbinate sample. According to the instructions for use (IFU), mid-turbinate swabs are required to be collected under medical supervision,13 which the CDC reinforces. There have been multiple studies that have demonstrated that mid-turbinate samples are effective for detection of other respiratory illnesses.14-17 Since mid-turbinate collection may have higher sensitivity than anterior nares or saliva testing, it is important to demonstrate that it can be safely collected without clinical supervision. Although some patients may be able to perform a mid-turbinate collection via a telehealth visit this would be a barrier to wide scale-up. Thus, the investigators will allow patients to self-collect a mid-turbinate sample with a collection swab. The swab will have an indicator line signaling the mean length to reach the mid-turbinate region in adults (approximately 1 inch, or 2 cms). The healthcare provider will then evaluate the patient for any adverse events related to the patient self-collection, such as pain and/or bleeding. If the incidence of adverse events is absent or very low (less than 5%) and the sensitivity of the mid-turbinate sample is superior to the anterior nares, patients could be allowed to sample their own mid-turbinate region without medical supervision. The proportion of participants experiencing each type of adverse event will be estimated along with a corresponding 95% exact confidence interval.

4.0 Summary The Covid-19 pandemic has created a global crisis that is affecting all sectors of society. To decrease the catastrophic economic and healthcare impacts of this virus, the availability of safe, inexpensive, and reliable testing will be necessary. This project aims to study the self-collection of a low-cost, rapid test (iAMP®) in three anatomic areas - the mid-turbinate, the nares and saliva - that, if validated, can help make widespread testing a real possibility. The secondary aim is to show that all of these areas can be safely self-collected without the need for clinician supervision. Decreasing barriers to Covid-19 testing and processing will help to mitigate this crisis and allow for a return to normal activities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 presenting for COVID-19 testing
* Subject able to tolerate nasopharyngeal swabs
* Subjects able to follow instructions for self-collection.

Exclusion Criteria:

* Subjects younger than 18
* Subjects unable to tolerate nasopharyngeal swabs
* Subjects unable to follow instructions
* Subjects unable or unwilling to provide informed consent and/or reliable contact information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SARS-CoV-2 positive and negative participants
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Validate iAMP testing kit | 1 month
  Validate the iAMP® testing kit for use in the mid-turbinate, anterior nares and with saliva collection and compare the sensitivities and specificities of each site to nasopharyngeal collection.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Felix, M.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Mooreland Reserve Health Center, New Berlin, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No